CLINICAL TRIAL: NCT03379402
Title: Utility of Sepsis-3 Definition, Causes and Factors Associated With Outcomes in Community-acquired Sepsis in Ubon Ratchathani, Northeast Thailand
Brief Title: Sepsis-3 Study in Northeast Thailand
Acronym: SEPSISIII
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Sanpasitthiprasong Hospital (Other Government); Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: HCR17001
Record Dates: First submitted 2017-12-04; First posted 2017-12-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Community-Acquired Infections
Keywords: causes of community-acquired sepsis; diagnostic tests
MeSH Terms: conditions — Sepsis; Community-Acquired Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Clinical specimens (including blood, urine, sputum, throat swabs and pus or wound swab) will be collected from each participant on admission for culture, PCR and serological tests, and other laboratory tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients presenting with sepsis: Adult patients, both males and females, presenting with sepsis will be approached for participation in the study.
  Interventions: Other: Specimens collection

INTERVENTIONS:
Other: Specimens collection — On admission: Blood samples 30.01 mL and other specimens (if available) for culture and other diagnostics tests including sputum, throat swab, urine (midstream urine), and pus which is part of routine practice for patients with sepsis at study site.
  Day 3: Blood (15 mL) for culture (10 mL) and PCR (5 mL). There will be no blood collection, if patient is discharged before day 3.

SUMMARY:
This is an observational study to evaluate the utility of the latest recommendation to define severity of infection for sepsis patients (sepsis-3), and to identify the aetiology and factors associated with outcome of community-acquired sepsis in Northeast Thailand.

Potential study participants will be adult patients who are presented at the hospital with community-acquired sepsis. Clinical specimens (including blood, urine, sputum, throat swabs and pus or wound swab) will be collected from each participant on admission for culture, PCR and serological tests, and other laboratory tests. Participants' treatment will be closely monitored during the duration of their hospital stay. Blood will be again collected at 72 hours after admission. Participants will be contacted at 28 days after admission to determine clinical outcome by phone interview with standardized script.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years old.
2. Thai nationality.
3. Required hospitalization as decided by the attending physician
4. Documented by attending physician that an infection is the primary cause of illness leading to the hospitalization. These can be infections due to any pathogens (bacteria, viruses, fungi and parasites).
5. qSOFA (quick Sepsis-related Organ Failure Assessment) score ≥ 2 defined as 2 or more of the following:

   * Respiratory rate ≥22 /min or required ventilator
   * Alteration of mental status (GCS<15 or 10T with endotracheal tube)
   * Systolic blood pressure ≤100 mm Hg

Exclusion Criteria:

1. Infection is not suspected to be a primary cause of the current illness episode leading to the hospitalization. For example, community-acquired sepsis is considered to be due to stroke, cardiovascular diseases, acute myocardial infarction, cancer, burn, injury, and trauma.
2. Hospitalized at the study site for this current episode for more than 24 hours before enrollment.
3. Hospitalized for this current episode for more than 72 hours at another primary/referring hospital
4. Prior to this current episode, the patient was admitted to any hospital within the last 30 days.
5. Prior to enrolment, it is documented by the attending physician that hospital acquired infection is associated with the cause of sepsis.

Please note that the following conditions are not exclusion criteria, and patients with the following conditions can be enrolled into the study.

* Confirmed diagnosis by any method of an infection as a major cause of illnesses leading to hospitalization. For example, a patient who already has had a definite diagnosis of malarial infection by blood smear.
* Clinical diagnosis of any specific disease or any specific syndromes such as acute infective diarrhea, acute pneumonia, acute encephalomyelitis and acute myocarditis.
* Suspected of having both infectious and non-infectious diseases and infectious disease is a primary cause of illnesses (primary diagnosis) leading to the hospitalization. For example, acute pneumonia with stroke as an underlying disease, etc.
* Patients who are admitted to other hospitals and referred to the study site. For example a referred patient who admit to the first hospital less than 24 hours prior to enrollment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients, both males and females, presenting with sepsis will be approached for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
28-day mortality after admission date | 2.5 years

SECONDARY OUTCOMES:
Causative organisms of community-acquired sepsis | 2.5 years
Respiration: Blood gas (PaO2 [mmHg]) | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Respiration: Type of oxygen support | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Respiration: FiO2 (% ) | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Respiration: SpO2 by pulse oximeter level (%) | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Coagulation: Platelet (per μL) | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Liver: Total Bilirubin (mg/dL) | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Cardiovascular: Mean Arterial Pressure (MAP) at enrolment (mmHg) | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Cardiovascular: Dosages (μg/kg/min) of inotropic | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Cardiovascular: Dosages (μg/kg/min) of vasopressor agents | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Central nervous system: Glasgow Coma Score | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Renal: Creatinine (mg/sdL) | 2.5 years
  Clinical parameters evaluated as according to Sepsis-3 guideline; Sequential Organ Failure Assessment (SOFA)
Hematology | 2.5 years
  Other laboratory measurement
Blood chemistry | 2.5 years
  Other laboratory measurement
Causes of sepsis associated with mortality outcome in patients with community-acquired sepsis in northeast Thailand | 2.5 years
Sepsis resuscitation associated with mortality outcome in patients with community-acquired sepsis in northeast Thailand | 2.5 years
Antimicrobial treatment associated with mortality outcome in patients with community-acquired sepsis in northeast Thailand | 2.5 years
Inflammatory associated with mortality outcome in patients with community-acquired sepsis in northeast Thailand | 2.5 years
Genetics factors with mortality outcome in patients with community-acquired sepsis in northeast Thailand | 2.5 years
Diagnostic tests for infection in community-acquired sepsis in NE Thailand | 2.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sappasithiprasong Hospital, Ubon Ratchathani, Thailand